CLINICAL TRIAL: NCT04183790
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Efficacy of ELX/TEZ/IVA Combination Therapy in Subjects With Cystic Fibrosis Who Are 6 Years of Age and Older
Brief Title: Evaluation of Long-term Safety and Efficacy of ELX/TEZ/IVA TC Combination Therapy in Participants With Cystic Fibrosis Who Are 6 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX19-445-107; 2019-001827-11 (EudraCT Number)
Expanded Access: NCT04702360 (Approved for marketing)
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants greater than or equal to (≥) 6 years and less than (<) 12 years of age and weighing <30 kilograms (kg) received ELX (elexacaftor) 100 milligram (mg) once daily (qd) /TEZ (tezacaftor) 50 mg qd/IVA (ivacaftor) 75 mg every 12 hours (q12h) and those weighing (≥) 30 kg received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg in the treatment period for up to 192 weeks. Participants ≥12 years of age received ELX 200 mg qd/ TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for up to 192 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Mono tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
The study evaluates the long-term safety, tolerability, efficacy, and pharmacodynamics of elexacaftor (ELX, VX-445) in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in participants with cystic fibrosis (CF).

ELIGIBILITY:
Key Inclusion Criteria:

* Completed study drug treatment in parent study (VX18-445-106 Part B, NCT03691779), or had study drug interruption(s) in parent study but completed study visits up to the last scheduled visit of the Treatment Period in the parent study

Key Exclusion Criteria:

* History of study drug intolerance in parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Northwell Health- Long Island Jewish Medical Center, New Hyde Park, New York
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia's Children's Hospital, Vancouver
- Ireland (2):
  - Children's Health Ireland at Crumlin, Dublin
  - Children's Health Ireland at Temple Street, Dublin
- United Kingdom (2):
  - Birmingham Children's Hospital - NHS Foundation Trust, Birmingham
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Wainwright C, McColley SA, McNally P, Powers M, Ratjen F, Rayment JH, Retsch-Bogart G, Roesch E, Ramsey B, McKone EF, Tullis E, Mall MA, Taylor-Cousar JL, Waltz D, Ahluwalia N, Chu C, Scirica CV, Davies JC. Long-Term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor in Children >/=6 Years with Cystic Fibrosis and at Least One F508del Allele: A 192-Week, Phase 3, Open-Label Extension Study. Am J Respir Crit Care Med. 2025 Oct;211(10):1915-1925. doi: 10.1164/rccm.202502-0512OC. PMID 40454869
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Wainwright C, McColley SA, McNally P, Powers M, Ratjen F, Rayment JH, Retsch-Bogart G, Roesch E, Ahluwalia N, Chin A, Chu C, Lu M, Menon P, Waltz D, Weinstock T, Zelazoski L, Davies JC. Long-Term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor in Children Aged ⩾6 Years with Cystic Fibrosis and at Least One F508del Allele: A Phase 3, Open-Label Clinical Trial. Am J Respir Crit Care Med. 2023 Jul 1;208(1):68-78. doi: 10.1164/rccm.202301-0021OC. PMID 37154609
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in two parts, Part A and Part B. Participants of both Parts A and B received the same treatment (ELX,TEZ,IVA). Therefore, results data were planned to be collected and analyzed for the overall population of the study and not for separate parts.
Pre-assignment Details: Participants from parent study VX18-445-106 Part B (NCT03691779) were enrolled in this study. A total of 64 participants were enrolled in this open label extension study.
Groups:
- Additional Participants for Cumulative Triple Combination (TC) Efficacy Set: This reporting arm represents the two additional participants in Cumulative TC Efficacy Set 106/107 from parent study 106 which were not enrolled in this study, but were included in the Cumulative TC efficacy 106/107 analysis set.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA | Additional Participants for Cumulative Triple Combination (TC) Efficacy Set
Started | 64 | 2
Part A Completed | 60 | 0
Rollover to Part B | 48 | 0
Cumulative TC Efficacy Set 106/107 | 64 (Cumulative TC Set includes participants who were enrolled and received at least 1 dose of study drug during the parent study (Study 106 Part B) and/or received at least 1 dose of study drug during this open label extension (OLE) study.) | 2 (Cumulative TC Set includes participants who were enrolled and received at least 1 dose of study drug during the parent study (Study 106 Part B) and/or received at least 1 dose of study drug during this open label extension (OLE) study. Two participants from parent study 106 Part B (not enrolled in this study) were included in this analysis set.)
Completed | 39 | 0
Not Completed | 25 | 2
Not completed — Participants did not rollover to Part B | 12 | 0
Not completed — Withdrawal of consent (not due to AE) | 6 | 0
Not completed — Commercial drug is available for participant | 6 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Not enrolled in 107 study | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug in this OLE study were included in the baseline characteristics.
Groups:
- ELX/TEZ/IVA: Participants ≥6 years and <12 years of age and weighing <30 kg received ELX 100 mg qd /TEZ 50 mg qd/IVA 75 mg q12h and those weighing ≥30 kg received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg in the treatment period for up to192 weeks. Participants ≥12 years of age received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for up to 192 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 56
  Not collected per local regulations | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55
  Asian | 0
  Not collected per local regulations | 8
  More than one Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Baseline up to Week 196
Population: OLE Safety Set was defined as all subjects who received at least 1 dose of study drug in this OLE study. Data for this outcome measure was planned to be collected and analyzed for the overall ELX/TEZ/IVA arm irrespective of Part A and B separately.
Measure: Count of Participants; unit: Participants
Groups:
- ELX/TEZ/IVA: Participants ≥6 years and <12 years of age and weighing <30kg received ELX 100 mg qd /TEZ 50 mg qd/IVA75 mg q12h and those weighing ≥30 kg received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg in the treatment period for up to 192 weeks. Participants ≥12 years of age received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for up to 192 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 64
Participants
  Participants with TEAEs | 64
  Participants with SAEs | 7

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline up to Week 192
Population: Open label Extension Full Analysis Set (OLE FAS) included all enrolled participants who have received at least 1 dose of study drug in the OLE study. Data for this outcome measure was planned to be collected and analyzed for the overall ELX/TEZ/IVA TC arm irrespective of Part A and B separately. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FEV1
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 27
percent predicted FEV1 | 9.6 [5.4 to 13.7]

3. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline up to Week 192
Population: OLE FAS. Data for this outcome measure was planned to be collected and analyzed for the overall ELX/TEZ/IVA TC arm irrespective of Part A and B separately. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 35
millimole per liter (mmol/L) | -57.9 [-63.3 to -52.5]

4. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 36
units on a scale | 10.0 [6.9 to 13.0]

5. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kg divided by squared height in meters (m^2).
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 39
kg/m^2 | 3.60 [2.98 to 4.23]

6. Secondary Outcome: Absolute Change in BMI-for-age Z-score
Description: BMI was defined as weight in kg divided by squared height in meters (m^2). The z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 39
z-score | 0.39 [0.19 to 0.59]

7. Secondary Outcome: Number of Participants With Pulmonary Exacerbations (PEx) for 106/107
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline up to Week 192
Population: The Cumulative TC Set includes participants who enrolled and received at least one dose of study drug during the parent study (445-106 Part B) and/or received at least one dose of study drug during this OLE Study. Data for this outcome measure was planned to be collected and analyzed for the overall ELX/TEZ/IVA TC arm irrespective of Part A and B separately. Here "Overall Number of Participants Analyzed" signifies those participants who evaluated for this specific outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 66
Participants | 9

8. Secondary Outcome: Number of CF-related Hospitalizations for 106/107
Description: The total number of CF related hospitalization (Planned + Unplanned) events across all participants were reported.
Time Frame: From Baseline up to Week 192
Population: The Cumulative TC Set. Data for this outcome measure was planned to be collected and analyzed for the overall ELX/TEZ/IVA TC arm irrespective of Part A and B separately. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this specific outcome measure.
Measure: Number; unit: hospitalizations
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 66
hospitalizations | 5

9. Secondary Outcome: Absolute Change in Lung Clearance Index 2.5 (LCI 2.5)
Description: The LCI2.5 index is the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting values and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured functional residual capacity (FRC). An LCI of 7.5 and below is normal; values greater than 7.5 are abnormal. LCI is able to detect abnormalities in lung function earlier than more traditional modalities such as spirometry.
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 25
index | -2.33 [-2.87 to -1.79]

10. Secondary Outcome: Absolute Change in Weight
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilogram (kg)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 39
Kilogram (kg) | 19.9 [18.1 to 21.7]

11. Secondary Outcome: Absolute Change in Weight-for-age Z-score
Description: The z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 39
z-score | 0.38 [0.20 to 0.55]

12. Secondary Outcome: Absolute Change in Height
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters (cm)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 39
centimeters (cm) | 23.1 [21.6 to 24.6]

13. Secondary Outcome: Absolute Change in Height-for-age Z-score
Description: as for outcome 11
Time Frame: From Baseline up to Week 192
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 39
z-score | 0.04 [-0.12 to 0.19]

ADVERSE EVENTS:
Time Frame: Day 1 Up to Week 196
Description: The OLE Safety Set is defined as all participants who received at least 1 dose of study drug in the OLE study.
Arm/Group | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 7/64
Other Adverse Events (participants affected / at risk) | 62/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=64)
Constipation (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2
Haematuria traumatic (Injury, poisoning and procedural complications) | 1
Idiopathic intracranial hypertension (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=64)
Ear pain (Ear and labyrinth disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 17
Fatigue (General disorders) | 10
Pyrexia (General disorders) | 28
COVID-19 (Infections and infestations) | 18
Ear infection (Infections and infestations) | 4
Hordeolum (Infections and infestations) | 9
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 8
Influenza (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 10
Pharyngitis streptococcal (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 19
Viral upper respiratory tract infection (Infections and infestations) | 7
Immunisation reaction (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 5
Bacterial test positive (Investigations) | 7
SARS-CoV-2 test positive (Investigations) | 8
Headache (Nervous system disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 40
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 21
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT04183790/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT04183790/SAP_001.pdf